CLINICAL TRIAL: NCT06806046
Title: A Phase 1, Open-label Study of Anti-CEACAM5 Antibody-Drug Conjugate Precemtabart Tocentecan (M9140) in Chinese Participants With Solid Tumors (PROCEADE-CRC-02)
Brief Title: Anti-CEACAM5 ADC Precemtabart Tocentecan (M9140) in Chinese Participants With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS202329_0003; CTR20244167 (Registry Identifier: China)
Record Dates: First submitted 2025-01-13; First posted 2025-02-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors; Colorectal Cancer
Keywords: ADC; Anti-CEACAM5; colorectal cancer; solid tumors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M9140 (Experimental)
  Interventions: Drug: M9140

INTERVENTIONS:
Drug: M9140 — M9140 will be administered every 3 weeks until progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study. There will be 2 dose levels, if the low dose level is tolerated, then M9140 will be escalated to the high dose level.
  Other Names: Precemtabart tocentecan

SUMMARY:
The purpose of this study is to evaluate the safety and early clinical activity of M9140 in Chinese participants with locally advanced or metastatic colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented histopathological diagnosis of locally advanced or metastatic CRC, who were intolerant/refractory to or progressed after standard systemic therapies for the advanced/metastatic stage that included and are restricted to a fluoropyrimidine, irinotecan, a platinum agent (e.g. oxaliplatin), an anti-EGFR agent (if clinically indicated, i.e. RAS/BRAF wt), and an anti-VEGF agent. Participants may have received previous treatment with trifluridine/tipiracil and/or regorafenib or fruquintinib, if locally indicated and available. Participants with a known MSI-H status must have received treatment with an immune checkpoint inhibitor (if locally indicated and available) unless contraindicated
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) below or equal to 1
* Participants with adequate hematologic, hepatic and renal function as defined in protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participant has a history of malignancy within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertropia, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years)
* Participants with known brain metastases, except those meeting the following criteria: Brain metastases that have been treated locally and are clinically stable for at least 4 weeks prior to the start of treatment; No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
* Participants with diarrhea (liquid stool) or ileus Grade > 1
* Cerebrovascular accident/stroke (< 6 months prior to enrollment)
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Up to 21 days (Each cycle is of 21 days)
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 8 months

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Plasma Concentrations of M9140 | Cycle 1 Day 1 (C1D1) - Predose, 6, 24, 168, 336 hr (hour) post dose: predose C2D1; C3D1 - Predose, 6, 24, 336 hr postdose; C4D1 - predose every 2 cycles until treatment discontinuation (20 months). [Each cycle is of 21 days]
Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment throughout the study duration until progressive disease or death up to approximately 8 months
Duration of Response (DoR) According to RECIST v1.1 as Assessed by Investigator | Time from first study treatment throughout the study duration until progressive disease or death up to approximately 8 months
Progression-free Survival (PFS) According to RECIST v1.1 | Time from first study treatment throughout the study duration until progressive disease or death up to approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202329_0003
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217341&parentIdentifier=MS202329_0003&attachmentIdentifier=1e49c0b6-fd7c-49cb-8e2b-e77dbf395055&fileName=CTR20244167_Details.pdf&versionIdentifier=